CLINICAL TRIAL: NCT02160782
Title: Long-Term, Open-Label Study With a Double-Blind, Placebo-Controlled, Randomized Drug Withdrawal Period of LUM001 (Maralixibat), an Apical Sodium-Dependent Bile Acid Transporter Inhibitor (ASBTi), in Patients With Alagille Syndrome
Brief Title: Safety and Efficacy Study of LUM001 (Maralixibat) With a Drug Withdrawal Period in Participants With Alagille Syndrome (ALGS)
Acronym: ICONIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUM001-304; 2013-005373-43 (EudraCT Number)
Expanded Access: NCT04530994 (Approved for marketing)
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome | interventions — maralixibat

STUDY DESIGN:
Intervention Model Description: Open-label single arm study with a randomized placebo-controlled parallel group period
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LUM001 (Maralixibat) (Experimental): LUM001, also known as Maralixibat (MRX) will be administered orally once a day (QD) up to 400 microgram per kilogram per day (mcg/kg/day) up to Week 52, followed by an increase in dose orally twice a day (BID) during long-term follow-up based on efficacy (serum bile acid [sBA] level and ItchRO[Obs] score) and safety assessment.
  Note: 400 mcg/kg maralixibat chloride is equivalent to 380 mcg/kg free maralixibat.
  Interventions: Drug: LUM001 (Maralixibat)
- Placebo (Placebo Comparator): Placebo will be administered orally once a day during randomized withdrawal period (Week 19 to Week 22)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LUM001 (Maralixibat) — LUM001, also known as Maralixibat (MRX) will be administered orally Once Daily (OD). To be administered Twice Daily (BID) for patients who are eligible.
  Arms: LUM001 (Maralixibat)
Drug: Placebo — Placebo will be administered orally once daily during randomized withdrawal period
  Arms: Placebo

SUMMARY:
This is a long-term, open-label study with a double-blind, placebo-controlled, randomized drug withdrawal period in children with Alagille Syndrome (ALGS) designed to evaluate the safety and efficacy of LUM001 (Also known as maralixibat or MRX).

DETAILED DESCRIPTION:
The study is divided into 6 parts: a 6-week open-label, dose escalation period, a 12-week open-label stable dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, a 26-week long-term stable dosing period, and an a 52-week optional follow-up treatment period, and a long-term optional follow-up treatment period for eligible participants who choose to stay on treatment with LUM001.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 12 months and 18 years inclusive.
* Diagnosis of ALGS.
* Evidence of cholestasis (one or more of the following):

  1. Total serum bile acid > 3x ULN for age.
  2. Conjugated bilirubin > 1 mg/dL.
  3. Fat soluble vitamin deficiency otherwise unexplainable.
  4. GGT > 3x ULN for age.
  5. Intractable pruritus explainable only by liver disease.
* Females of childbearing potential must have a negative serum pregnancy test during Screening.
* Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial.
* Participant is expected to have a consistent caregiver(s) for the duration of the study.
* Informed consent and assent (per IRB/IEC) as appropriate.
* Access to phone for scheduled calls from study site.
* Caregivers (and age-appropriate participants) must be willing and able to use an eDiary device during the study.
* Caregivers (and age-appropriate participants) must digitally accept the licensing agreement in the eDiary software.
* Caregivers (and age-appropriate participants) must complete at least 10 eDiary reports (morning or evening) during each of two consecutive weeks of the screening period (maximum possible reports = 14 per week).
* Average daily score >2 on the Itch Reported Outcome (ItchRO™) questionnaire (maximum possible daily score of 4) for two consecutive weeks in the screening period, prior to dosing. A daily score is the higher of the scores for the morning and evening ItchRO. The average daily score is the sum of all daily scores divided by the number of days the ItchRO was completed.

Inclusion Criteria for participants to be eligible for the 52-week optional follow-up treatment period:

* Completed the protocol through the Week 48 visit with no safety concerns. Participants who were discontinued due to safety reasons can be rechallenged if blood tests are back to relatively normal values for this patient population and participant does not meet any of the protocol's stopping rules. The decision will be made by the investigator in consultation with the sponsor medical monitor.
* Participants who have undergone a surgical disruption of the enterohepatic circulation will not be eligible to enter into the follow up treatment period.
* Participants who were discontinued for other reasons will be considered for the 52-week optional follow-up treatment period on an individual basis. The decision will be made by the investigator in consultation with the sponsor medical monitor.

Inclusion Criteria for participants with LUM001dosing interruption <7 days, or >=7 days:

* The Participant has either: completed the protocol through the Week 48 visit with no major safety concerns OR discontinued due to safety reasons judged unrelated to the study drug, and laboratory results have returned to levels acceptable for this patient population or individual and participant does not meet any of the protocol's stopping rules at the time of entry into the follow-up period. The decision will be made by the investigator in consultation with the sponsor medical monitor. [Participants who were discontinued for other reasons will be considered on an individual basis.]
* Females of childbearing potential must have a negative urine or serum pregnancy test (beta- human chorionic gonadotropin [β-hCG]) at the time of entry into the long-term optional follow-up treatment period.
* Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial.
* Informed consent and assent (per IRB/EC) as appropriate.
* Access to phone for scheduled calls from study site.
* Caregivers (and age-appropriate participants) must be willing and able to use an eDiary device during the study.

Exclusion Criteria:

* Chronic diarrhea requiring ongoing intravenous fluid or nutritional intervention.
* Surgical interruption of the enterohepatic circulation.
* Previous liver transplant
* Decompensated cirrhosis (ALT >15 x ULN, INR >1.5 [unresponsive to vitamin K therapy], albumin <3.0 g/dL, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy).
* History or presence of other concomitant liver disease.
* History or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (eg, inflammatory bowel disease).
* History or presence of gallstones or kidney stones.
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Cancers, except for in situ carcinoma, or cancers treated at least 5 years prior to Screening with no evidence of recurrence.
* Recent medical history or current status that suggests that the participant may be unable to complete the study.
* Any female who is pregnant or lactating or who is planning to become pregnant during the study period.
* Known history of alcohol or substance abuse.
* Administration of bile acid or lipid binding resins within 28 days prior to screening and throughout the trial.
* Known hypersensitivity to LUM001 or any of its components.
* Receipt of investigational drug, biologic, or medical device within 28 days prior to screening, or 5 half-lives of the study agent, whichever is longer.
* History of non-adherence to medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to nonadherence with the study protocol based upon investigator judgment.
* Any other conditions or abnormalities which, in the opinion of the investigator or sponsor medical monitor, may compromise the safety of the participant, or interfere with the participant participating in or completing the study.
* Participants weighing over 50 kg at screening.

Exclusion Criteria for participants with LUM001 dosing interruption >=7 days:

- All exclusion criteria mentioned above apply upon entry into the long-term optional follow-up period, with the exception of participants weighing over 50 kg at screening.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (9):
- Australia (2):
  - Children's Hospital Westmead, Westmead, New South Wales
  - The Royal Children's Hospital Melbourne, Parkville, Victoria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (3):
  - Hopital Femme Mere Enfant De Lyon, Bron
  - Hopital Necker-Enfants Malades, Paris
  - Hopital Kremlin Bicetre, Paris
- The Children's Memorial Health Institute, Warsaw, Poland
- Hospital Universitario La Paz- Hospital Materno Infantil, Madrid, Spain
- Paediatric Liver Center, Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamath BM, Goldstein A, Howard R, Garner W, Vig P, Marden JR, Billmyer E, Anderson A, Kirson N, Jacquemin E, Gonzales E. Maralixibat Treatment Response in Alagille Syndrome is Associated with Improved Health-Related Quality of Life. J Pediatr. 2023 Jan;252:68-75.e5. doi: 10.1016/j.jpeds.2022.09.001. Epub 2022 Sep 10. PMID 36096175
- [Derived] Gonzales E, Hardikar W, Stormon M, Baker A, Hierro L, Gliwicz D, Lacaille F, Lachaux A, Sturm E, Setchell KDR, Kennedy C, Dorenbaum A, Steinmetz J, Desai NK, Wardle AJ, Garner W, Vig P, Jaecklin T, Sokal EM, Jacquemin E. Efficacy and safety of maralixibat treatment in patients with Alagille syndrome and cholestatic pruritus (ICONIC): a randomised phase 2 study. Lancet. 2021 Oct 30;398(10311):1581-1592. doi: 10.1016/S0140-6736(21)01256-3. Epub 2021 Oct 28. PMID 34755627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were enrolled at 9 sites in 6 countries (Australia, UK, France, Poland, Spain and Belgium) between 28 October 2014 and 11 September 2015
Pre-assignment Details: A total of 36 patients were screened for the study. 31 patients were enrolled, while 5 patients were screen failures.
Groups:
- Open-label Period: Maralixibat (LUM001): All participants received Maralixibat (LUM001:MRX) at doses of up to 400 μg/kg once daily (QD) during a 6-week open-label dose-escalation period, followed by a 12-week open-label stable-dosing period. All participants reached 400 μg/kg QD for this period.
  Participants were randomized 1:1 to continue to receive MRX or placebo (Pbo) for 4 weeks between the start of Week 19 and the end of Week 22 (the double-blind, placebo-controlled study drug withdrawal period).
  All participants, caregivers, monitors, and study center personnel related to the study, except for the central pharmacist who prepared the study drug, were blinded to the participants' study drug withdrawal period treatment assignment during the randomized withdrawal (RWD) period.
  Participants who received placebo during the RWD period returned to MRX 400 μg/kg QD in a 26-week long-term exposure period to complete 48 weeks of treatment.
  Participants who received MRX during the RWD period continued in a 26-week long-term exposure period to complete 48 weeks of treatment.
- Randomized Withdrawal Period: MRX: Participants continued to receive MRX at 400 μg/kg QD during the RWD period
- Randomized Withdrawal Period: Placebo: Participants received a corresponding placebo during the RWD period
- After Randomized Withdrawal Period: Maralixibat: Participants who received placebo during the RWD period returned to the MRX 400 μg/kg QD in a 26-week long-term exposure period to complete 48 weeks of treatment. Participants who received MRX during the RWD period continued in a 26-week long-term exposure period to complete 48 weeks of treatment. Participants remained blinded to their assigned arm during the RWD period.
- Long-term Extension Period: Maralixibat: The long-term extension (LTE) period consisted of 2 phases: (1) a 52-week optional follow-up treatment period (Weeks 49-100), during which participants received up to 400 μg/kg QD MRX. This was followed by: (2) a long-term optional follow-up treatment period (>Week 100) during which participants received up to 400 μg/kg BID doses of MRX.
Period: Open-label Period: Maralixibat
Arm/Group | Open-label Period: Maralixibat (LUM001) | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo | After Randomized Withdrawal Period: Maralixibat | Long-term Extension Period: Maralixibat
Started | 31 | 0 | 0 | 0 | 0
Completed | 29 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Period: Randomized Withdrawal Period- Pbo vs MRX
Arm/Group | Open-label Period: Maralixibat (LUM001) | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo | After Randomized Withdrawal Period: Maralixibat | Long-term Extension Period: Maralixibat
Started | 0 | 13 | 16 | 0 | 0
Completed | 0 | 13 | 16 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: After Randomized Withdrawal: Maralixibat
Arm/Group | Open-label Period: Maralixibat (LUM001) | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo | After Randomized Withdrawal Period: Maralixibat | Long-term Extension Period: Maralixibat
Started | 0 | 0 | 0 | 29 | 0
Completed | 0 | 0 | 0 | 23 | 0
Not Completed | 0 | 0 | 0 | 6 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Did not consent to protocol amendment for long term extension | 0 | 0 | 0 | 5 | 0
Period: Long-term Extension Period: Maralixibat
Arm/Group | Open-label Period: Maralixibat (LUM001) | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo | After Randomized Withdrawal Period: Maralixibat | Long-term Extension Period: Maralixibat
Started | 0 | 0 | 0 | 0 | 23
Completed | 0 | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 0 | 9
Not completed — Did not consent to protocol amendment | 0 | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by caregiver | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label Period: Maralixibat: All participants received MRX at doses of up to 400 μg/kg once daily (QD) during a 6-week open-label dose-escalation period, followed by a 12-week open-label stable-dosing period. All participants reached 400 μg/kg QD for this period.
Arm/Group | Open-label Period: Maralixibat
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years of age] | 5.4 (4.25)
Age, Customized [Count of Participants; unit: Participants]
  <2 years | 6
  2 to 4 years | 9
  5 to 8 years | 9
  9 to 12 years | 4
  13 to 18 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not collected.
  Asian | NA — Not collected.
  Native Hawaiian or Other Pacific Islander | NA — Not collected.
  Black or African American | NA — Not collected.
  White | NA — Not collected.
  More than one race | NA — Not collected.
  Unknown or Not Reported | NA — Not collected.
Region of Enrollment [Number; unit: participants]
  Australia | 9
  Belgium | 5
  France | 9
  Poland | 3
  Spain | 2
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 18 to Week 22 in Fasting sBA Levels in Participants Who Had a Reduction in sBA ≥50% From Baseline to Week 12 or Week 18
Description: The primary efficacy endpoint of this study was the mean change from Week 18 to Week 22 (the RWD period) of fasting sBA levels in participants who had a reduction in sBA ≥50% from baseline to Week 12 or Week 18 (Modified Intent-to-Treat [MITT] Population). Five participants in the MRX group and 10 participants in the placebo group met the prespecified sBA reduction criteria.
Time Frame: Week 18 to Week 22
Population: Primary outcome used the (Modified Intent-to-Treat [MITT]Population. The MITT population is defined as participants who had a reduction in sBA ≥50% from baseline to Week 12 or Week 18. Five participants in the MRX group and 10 participants in the placebo group met the prespecified sBA reduction criteria.
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 5 | 10
μmol/L | -21.73 (43.125) | 95.55 (30.488)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in fasting sBA levels was evaluated using an analysis of covariance (ANCOVA) model with treatment group as a factor, and Week 18 sBA as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the MITT population, which included all participants who were enrolled, received study drug through Week 18, and had a reduction from baseline in sBA of ≥50% at the Week 12 or Week 18 measurement; Test type: Equivalence — The P-value for testing if the treatment group least squares (LS) means were equal was calculated to determine if the change in sBA levels between the treatment groups was statistically significant; p = 0.0464, ANCOVA; Mean Difference (Net) = -117.28, 95% CI 2-sided [-232.38 to -2.18], Standard Error of Mean 52.828

2. Secondary Outcome: Change From Baseline to Week 18 in Fasting sBA Levels
Description: This secondary efficacy endpoint is the mean change from baseline to Week 18 in fasting sBA levels
Time Frame: Baseline to Week 18
Population: Values were collected from 31 participants at baseline. Values were collected at Week 18 from 29 of the 31 participants who contributed values at baseline.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- Open-label Period: MRX Baseline; Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in fasting sBA levels
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 29
μmol/L | 283.43 (210.569) | 192.50 (161.278)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; This analysis investigated whether a statistically significant change in sBA levels was observed when comparing baseline to Week 18 (the open-label period, during which all participants received MRX). The analysis was based on the ITT population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in sBA levels between baseline and Week 18 (the open-label period) was statistically significant; p = 0.0005, Student's t-test — Data for this analysis were obtained from 31 participants at baseline; 29 of those participants contributed Week 18 data; Mean Difference (Net) = -87.73, 95% CI 2-sided [-133.37 to -42.09], Standard Deviation 119.979

3. Secondary Outcome: Change From Baseline to Week 18 in Pruritus as Measured by ItchRO (Obs)
Description: This secondary efficacy endpoint is the change from baseline to Week 18 in pruritus as measured by ItchRO(Obs) weekly average morning score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe).
Time Frame: Baseline to Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Open-label Period: MRX Baseline; Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in ItchRO(Obs) and ItchRO(Pt)
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 29
Points | 2.909 (0.5480) | 1.203 (0.8446)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; This analysis investigated whether a statistically significant change in ItchRO(Obs) score was observed when comparing baseline to Week 18 (the open-label period, during which all participants received MRX). The analysis was based on the ITT population. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ItchRO(Obs) scores between baseline and Week 18 (the open-label period) was statistically significant; p < 0.0001, Student's t-test; Mean Difference (Net) = -1.704, 95% CI 2-sided [-2.051 to -1.357], Standard Deviation 0.9114

4. Secondary Outcome: Change From Baseline to Week 18 in Pruritus as Measured by ItchRO (Pt)
Description: This secondary efficacy endpoint is the change from baseline to Week 18 in pruritus as measured by ItchRO(Pt) weekly average morning score
Time Frame: Baseline to Week 18
Population: NOTE: 2 participants discontinued prior week 18 and did not provide data.
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Open-label Period: MRX Baseline; Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in ItchRO(Pt)
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 29
Points | 2.903 (0.6616) | 0.831 (0.8122)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; This analysis investigated whether a statistically significant change in ItchRO(Pt) score was observed when comparing baseline to Week 18 (the open-label period, during which all participants received MRX). The analysis was based on the ITT population. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ItchRO(Pt) scores between baseline and Week 18 (the open-label period) was statistically significant; p < 0.0001, Student's t-test; Mean Difference (Net) = -2.072, 95% CI 2-sided [-2.645 to -1.498], Standard Deviation 0.9931

5. Secondary Outcome: Change From Week 18 to Week 22 in Pruritus as Measured by ItchRO(Obs)
Description: This secondary efficacy endpoint is the change from Week 18 to Week 22 in pruritus as measured by ItchRO(Obs) weekly average morning score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe).
Time Frame: Week 18 to Week 22
Population: For Maralixibat, n=12 for ItchRO(Obs) weekly average morning score For Placebo, n=16 for ItchRO(Obs) weekly average morning score
Measure: Least Squares Mean (Standard Error); unit: Points
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 12 | 16
Points | 0.217 (0.2345) | 1.700 (0.2031)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in ItchRO(Obs) was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 ItchRO(Obs) as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug; Test type: Equivalence — The P-value for testing if the treatment group LS means were equal was calculated to determine if the change in ItchRO(Obs) between the treatment groups was statistically significant; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.483, 95% CI 2-sided [-2.122 to -0.844], Standard Error of Mean 0.3103

6. Secondary Outcome: Change From Week 18 to Week 22 in Pruritus as Measured by ItchRO(Pt)
Description: This secondary efficacy endpoint is the change from Week 18 to Week 22 in pruritus as measured by ItchRO(Pt) weekly average morning score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe).
Time Frame: Week 18 to Week 22
Population: ItchRO(Pt) was completed independently in participants 9 years old or older. Children between the ages of 5 and 8 years old completed the patient instrument with the assistance of their caregiver, if needed.
Measure: Least Squares Mean (Standard Error); unit: Points
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 5 | 9
Points | -0.149 (0.3719) | 1.839 (0.2771)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in ItchRO (Pt) was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 ItchRO(Pt) as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug; Test type: Equivalence — The P-value for testing if the treatment group LS means were equal was calculated to determine if the change in ItchRO(Pt) between the treatment groups was statistically significant. While the number of participants included in analysis for the end point indicates 28, there were only 14; n = 5 for ItchRO(Pt): MRX and n = 9 for ItchRO(Pt): placebo; p = 0.0013, ANCOVA; Mean Difference (Net) = -1.988, 95% CI 2-sided [-3.009 to -0.967], Standard Error of Mean 0.4641

7. Secondary Outcome: Change From Baseline to Week 18 in Alkaline Phosphatase
Description: This secondary efficacy endpoint is the mean change from baseline to Week 18 in ALP
Time Frame: Baseline to Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Open-label Period: MRX Baseline: This secondary efficacy endpoint is the mean change from baseline to Week 18 in fasting ALP levels
- Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in ALP levels
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 29
U/L | 601.3 (274.77) | 580.8 (215.50)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; This analysis investigated whether a statistically significant change in ALP levels was observed when comparing baseline to Week 18 (the open-label period, during which all participants received MRX). The analysis was based on the ITT population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ALP levels between baseline and Week 18 (the open-label period) was statistically significant; p = 0.2163, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -27.8, 95% CI 2-sided [-72.8 to 17.2], Standard Deviation 118.33

8. Secondary Outcome: Change From Week 18 to Week 22 in Alkaline Phosphatase
Description: This secondary efficacy endpoint is the mean change from Week 18 to Week 22 in ALP
Time Frame: Week 18 to Week 22
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 13 | 16
U/L | 2.8 (22.55) | -7.2 (20.31)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in ALP levels was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 ALP as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug; Test type: Equivalence — The P-value for testing if the treatment group LS means were equal was calculated to determine if the change in ALP levels between the treatment groups was statistically significant; p = 0.7455, ANCOVA; Mean Difference (Net) = 10, 95% CI 2-sided [-52.6 to 72.6], Standard Error of Mean 30.44

9. Secondary Outcome: Change From Baseline to Week 18 in Alanine Aminotransferase
Description: This secondary efficacy endpoint is the mean change from baseline to Week 18 in ALT
Time Frame: Baseline to Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Open-label Period: MRX Baseline; Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in ALT levels
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 29
U/L | 181.0 (108.56) | 177.4 (92.08)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; This analysis investigated whether a statistically significant change in ALT levels was observed when comparing baseline to Week 18 (the open-label period, during which all participants received MRX). The analysis was based on the ITT population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ALT levels between baseline and Week 18 (the open-label period) was statistically significant; p = 0.9358, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.3, 95% CI 2-sided [-33.4 to 30.9], Standard Deviation 84.54

10. Secondary Outcome: Change From Week 18 to Week 22 in Alanine Aminotransferase
Description: This secondary efficacy endpoint is the mean change from Week 18 to Week 22 in alanine aminotransferase (ALT)
Time Frame: Week 18 to Week 22
Population: The difference between treatment groups in change from Week 18 to Week 22 in ALT levels was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 ALT as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 13 | 16
U/L | 34.5 (14.04) | 19.4 (12.56)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in ALT levels was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 ALT as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug; Test type: Equivalence — The P-value for testing if the treatment group LS means were equal was calculated to determine if the change in ALT levels between the treatment groups was statistically significant; p = 0.4472, ANCOVA; Mean Difference (Net) = 15.1, 95% CI 2-sided [-25.1 to 55.2], Standard Error of Mean 19.53

11. Secondary Outcome: Change From Baseline to Week 18 in Total Bilirubin
Description: This secondary efficacy endpoint is the mean change from baseline to Week 18 in total bilirubin
Time Frame: Baseline to Week 18
Population: Open-label period: MRX baseline v Open-label period: MRX Week 18
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Open-label Period: MRX Baseline; Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in total bilirubin
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 29
mg/dL | 6.09 (5.781) | 5.12 (5.337)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in total bilirubin levels between baseline and Week 18 (the open-label period) was statistically significant; p = 0.0893, Student's t-test; Mean Difference (Net) = -0.47, 95% CI 2-sided [-1.01 to 0.08], Standard Deviation 1.424

12. Secondary Outcome: Change From Week 18 to Week 22 in Total Bilirubin
Description: This secondary efficacy endpoint is the mean change from Week 18 to Week 22 in total bilirubin
Time Frame: Week 18 to Week 22
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 13 | 16
mg/dL | 0.32 (0.265) | 0.46 (0.238)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in total bilirubin was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 total bilirubin as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug; Test type: Equivalence — The P-value for testing if the treatment group LS means were equal was calculated to determine if the change in total bilirubin between the treatment groups was statistically significant; p = 0.7, ANCOVA; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.88 to 0.6], Standard Error of Mean 0.361

13. Secondary Outcome: Change From Baseline to Week 18 in Direct Bilirubin
Description: This secondary efficacy endpoint is the mean change from baseline to Week 18 in direct bilirubin
Time Frame: Baseline to Week 18
Population: Values from the open-label period were collected from 31 participants at baseline. Values were collected at Week 18 from 28 of the 31 participants who contributed values at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Open-label Period: MRX Baseline; Open-label Period: MRX Week 18: This secondary efficacy endpoint is the mean change from baseline to Week 18 in direct bilirubin
Arm/Group | Open-label Period: MRX Baseline | Open-label Period: MRX Week 18
Number analyzed (Participants) | 31 | 28
mg/dL | 4.57 (3.666) | 3.98 (3.369)
Statistical Analysis 1: Comparison: Open-label Period: MRX Baseline vs Open-label Period: MRX Week 18; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in direct bilirubin levels between baseline and Week 18 (the open-label period) was statistically significant; p = 0.0139, Student's t-test; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.9 to -0.11], Standard Deviation 1.012

14. Secondary Outcome: Change From Week 18 to Week 22 in Direct Bilirubin
Description: This secondary efficacy endpoint is the mean change from Week 18 to Week 22 in direct bilirubin
Time Frame: Week 18 to Week 22
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 12 | 15
mg/dL | 0.13 (0.195) | 0.14 (0.174)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: MRX vs Randomized Withdrawal Period: Placebo; The difference between treatment groups in change from Week 18 to Week 22 in direct bilirubin levels was evaluated using an ANCOVA model with treatment group as a factor, and Week 18 direct bilirubin as a covariate. The analysis used a tabulation of fitted summary statistics from ANCOVA in the intent-to-treat population, which included all participants who were enrolled, and received at least one dose of study drug; Test type: Equivalence — The P-value for testing if the treatment group LS means were equal was calculated to determine if the change in direct bilirubin between the treatment groups was statistically significant; p = 0.9517, ANCOVA; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.56 to 0.53], Standard Error of Mean 0.265

ADVERSE EVENTS:
Time Frame: Baseline to study completion (median of 2 years)
Description: All treatment-emergent AEs, whether observed by the Investigator, reported by the participant, the participant's caregiver, from laboratory findings, or other means, were recorded on the AE eCRF and medical record. 'Occurrences' relates to the number of events; 'subjects affected' relates to the number of participants who experienced the AE.
Groups:
- Open-label Period: Maralixibat (LUM001): All participants received MRX at doses of up to 400 μg/kg once daily (QD) during a 6-week open-label dose-escalation period, followed by a 12-week open-label stable-dosing period. All participants reached 400 μg/kg QD for this period.
- Safety Population: The safety population was defined as all participants who were assigned and received at least one dose of the study drug.
Arm/Group | Open-label Period: Maralixibat (LUM001) | Randomized Withdrawal Period: MRX | Randomized Withdrawal Period: Placebo | After Randomized Withdrawal Period: Maralixibat | Long-term Extension Period: Maralixibat | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/13 | 0/16 | 0/29 | 0/23 | 0/31
Serious Adverse Events (participants affected / at risk) | 4/31 | 1/13 | 1/16 | 5/29 | 6/23 | 13/31
Other Adverse Events (participants affected / at risk) | 29/31 | 7/13 | 12/16 | 25/29 | 23/23 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Period: Maralixibat (LUM001) (N=31) | Randomized Withdrawal Period: MRX (N=13) | Randomized Withdrawal Period: Placebo (N=16) | After Randomized Withdrawal Period: Maralixibat (N=29) | Long-term Extension Period: Maralixibat (N=23) | Safety Population (N=31)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Marrow hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Period: Maralixibat (LUM001) (N=31) | Randomized Withdrawal Period: MRX (N=13) | Randomized Withdrawal Period: Placebo (N=16) | After Randomized Withdrawal Period: Maralixibat (N=29) | Long-term Extension Period: Maralixibat (N=23) | Safety Population (N=31)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (4)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Pyrexia (General disorders) | 6 (12) | 0 (0) | 1 (1) | 7 (12) | 10 (27) | 17 (52)
Breath holding (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychological trauma (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (7) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 6 (12)
Head injury (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 3 (8)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (5)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Vitamin A increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 8 (12) | 13 (18)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 7 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (4) | 4 (10) | 9 (19)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 3 (6)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (22) | 1 (1) | 1 (1) | 6 (12) | 12 (31) | 18 (67)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (18) | 1 (1) | 1 (1) | 5 (10) | 7 (18) | 18 (48)
Faeces pale (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lip discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (8)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (15) | 1 (1) | 1 (2) | 2 (3) | 8 (13) | 16 (34)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 5 (5) | 2 (3) | 0 (0) | 9 (13)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligamentitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitamin A deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin C deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 3 (7)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 4 (4) | 5 (6) | 8 (14)
Epstein-Barr virus infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (7) | 7 (9)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (6)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 8 (21) | 9 (46) | 13 (73)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (3) | 0 (0) | 3 (3) | 4 (6) | 9 (28)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 8 (8)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analyzed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02160782/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02160782/SAP_001.pdf